CLINICAL TRIAL: NCT06541613
Title: Bilateral External Oblique Intercostal Plane Block (EOIPB) an Alternative Analgesic Technique in Patients Scheduled for Laparoscopic Cholecystectomy: A Randomized Controlled Study
Brief Title: Bilateral External Oblique Intercostal Plane Block in Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Moshira sayed mohamed, Assistant lecturer, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PT (831)
Record Dates: First submitted 2024-07-21; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: External Oblique Intercostal Plane Block; Laparoscopic Cholecystectomy
Keywords: EOIPB, alternative analgesic, laparoscopic cholecystectomy
MeSH Terms: interventions — Anesthetics, Local; Bupivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: 38 patients will be enrolled in the study and divided into two groups either (EOIPB group (E) or Control group (C). Randomization will be done by allocation 1:1 of scheduled cases per day.
Who Masked: Participant, Care Provider, Investigator
Masking Description: the investigator responsible for block administration will not be aware of the content of the medications prepared whether they are the local anesthetics or normal saline. also the patients will not be aware of the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- The EOIPB ( E) group (Experimental): EOIPB will be administered by a single anesthetists following the intubation. A linear ultrasound transducer is positioned in the sagittal plane at the 6th rib level, between the anterior axillary and midclavicular lines. The ribs, lungs, pleura, intercostal muscles, external oblique muscle and subcutaneous tissue are visualized in the image. The in-plane technique with a 22G, 80 mm block needle is used to inject 30 ml of 0.25% bupivacaine into the external oblique intercostal plane on both sides.
  Interventions: Drug: local anesthetic injection (bupivacaine)
- The Control Group (C) (Placebo Comparator): Control group of patients will receive standard multimodal analgesia. Using us guidance, the external oblique intercostal plane is identified and 30 ml normal saline instead of LA will be injected in the control group.
  Interventions: Other: normal saline injection

INTERVENTIONS:
Drug: local anesthetic injection (bupivacaine) — The in-plane technique with a 22G, 80 mm block needle is used to inject 30 ml of 0.25% bupivacaine into the external oblique intercostal plane on both sides.
  Other Names: bupivacaine
  Arms: The EOIPB ( E) group
Other: normal saline injection — the control group will receive 30ml of normal saline bilaterally into the external oblique intercostal plane on both sides
  Other Names: Placebo
  Arms: The Control Group (C)

SUMMARY:
Pain after laparoscopic cholecystectomy (LC) is a common complaint that prolongs hospital stay and thus increases morbidity. There are three primary sources of pain after LC, incision site, local and systemic effects of pneumoperitoneum, and post cholecystectomy wound to the liver. External oblique intercostal plane block (EOIPB) has recently been described as a novel block for upper abdomen surgery. the probable mechanism of the block with the dyeing of both the anterior and lateral branches of the intercostal nerves T7-T10. This block also provides a dermatomal sensory block at the T6-T10 level in the anterior axillary region and the T6-T9 level in the midline.

DETAILED DESCRIPTION:
EOIPB has the benefit of being performed with the patient supine when compared with QLB and ESPB. It also has an advantage over SIPB in that it produces greater analgesia throughout the midline of the abdomen. The hypothesis of this randomized study is that patients who will undergo EOIPB will have lower opioid consumption in the postoperative period than patients who receive routine multimodal analgesia alone. The study aims to assess pain control in the immediate postoperative period by assessment of Numerical Rating scale (NRS), time for the first analgesic request as well as total morphine intake in the first 24 hours after surgery.

Study design:

This is a prospective, randomized double blinded control study which will be conducted in department of anesthesia and surgical Intensive care unit at Theodor Bilharz Research Institute after approval by research ethics committee and patient informed consent. 50 patients will be enrolled in the study and divided into two groups either (EOIPB group (E) or Control group (C). Randomization will be done by allocation 1:1 of scheduled cases per day.

Sample size: 38 patients

ELIGIBILITY:
Inclusion Criteria:

1. ASA 1-2.
2. Patients undergoing elective laparoscopic cholecystectomy with estimated pneumoperitoneum time of 60 to 90 min.-

Exclusion Criteria:

1. Coagulation disorders.
2. Liver/ kidney disease
3. Previous abdominal surgery
4. Infection in the block site
5. Chronic opioid use
6. Local anesthetic (LA) allergy,
7. Pregnancy, or BMI ≥35 kg/m2
8. Duration of surgery (≥ 2.5 h due to surgical complications), -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
total morphine consumption | the first 24 hours postoperatively
  the total analgesic (morphine) requirements in the first 24 hours postoperatively will be calculated

SECONDARY OUTCOMES:
NRS | 6 hours postoperatively
  Numerical rating scale for pain recorded at 15,30, 60 minutes postopetaively.

CONTACTS AND LOCATIONS:
Overall Officials: Moshira Amer, M.D., Principal Investigator — Theodor Bilharz Research Institute
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
the data of the participants will be available upon request from the principal investigator.

REFERENCES:
- [Background] Selvi O, Tulgar S, Senturk O, Serifsoy TE, Thomas DT, Deveci U, Ozer Z. Is a Combination of the Serratus Intercostal Plane Block and Rectus Sheath Block Superior to the Bilateral Oblique Subcostal Transversus Abdominis Plane Block in Laparoscopic Cholecystectomy? Eurasian J Med. 2020 Feb;52(1):34-37. doi: 10.5152/eurasianjmed.2019.19048. PMID 32158311
- [Background] Hamilton DL, Manickam BP, Wilson MAJ, Abdel Meguid E. External oblique fascial plane block. Reg Anesth Pain Med. 2019 Jan 11:rapm-2018-100256. doi: 10.1136/rapm-2018-100256. Online ahead of print. No abstract available. PMID 30635518
- [Background] White L, Ji A. External oblique intercostal plane block for upper abdominal surgery: use in obese patients. Br J Anaesth. 2022 May;128(5):e295-e297. doi: 10.1016/j.bja.2022.02.011. Epub 2022 Mar 3. No abstract available. PMID 35249704